CLINICAL TRIAL: NCT02883829
Title: Health Promotion in Transition: Effects of Web-Based Health Information on Disease Management and Risk Behavior for Youth With Type 1 Diabetes in College
Brief Title: Effects of Web-Based Health Information on Risk Behavior for Youth With Type 1 Diabetes in College
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Elissa R. Weitzman, Associate Scientist, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-P00023029
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer-Based Delivery (Experimental): The Peer-Based Delivery Arm will receive a brief health information intervention (delivered as video content) about diabetes self-management and alcohol use risks, measuring effects on health knowledge. For this arm, a peer will be the spokesperson delivering the intervention content.
  Interventions: Behavioral: Peer-Based Web-Based Health Information
- Provider-Based Delivery (Experimental): The Provider-Based Delivery Arm will receive a brief health information intervention (delivered as video content) about diabetes self-management and alcohol use risks, measuring effects on health knowledge. For this arm, a healthcare provider will be the spokesperson delivering the intervention content.
  Interventions: Behavioral: Provider-Based Web-Based Health Information

INTERVENTIONS:
Behavioral: Peer-Based Web-Based Health Information — The intervention will be a brief vignette to present educational content about alcohol use risks for Type 1 Diabetes; framed and delivered from a peer-based source. The content for the intervention will be drawn on existing theories of behavior change, including the concepts of 'consciousness raising', 'self-reevaluation' and 'helping relationships'. The intervention will comprise of PowerPoint slides for final implementation as a narrated video that can be posted to a website for participant viewing.
  Arms: Peer-Based Delivery
Behavioral: Provider-Based Web-Based Health Information — The intervention will be a brief vignette to present educational content about alcohol use risks for Type 1 Diabetes; framed and delivered from a provider-based source. The content for the intervention will be drawn on existing theories of behavior change, including the concepts of 'consciousness raising', 'self-reevaluation' and 'helping relationships'. The intervention will comprise of PowerPoint slides for final implementation as a narrated video that can be posted to a website for participant viewing.
  Arms: Provider-Based Delivery

SUMMARY:
Adolescence and emerging adulthood are critical periods during which health outcomes may be imperiled for youth with Type 1 Diabetes (T1D). Due to the strong presence of alcohol use in the college environment, college students with T1D may be especially vulnerable to these risks.

Our goal is to develop preliminary evidence in support of a scalable intervention targeting diabetes health management and alcohol use avoidance for college youth with T1D. For this project the investigators will engage at least 120 youth with T1D in college. The study sample will be drawn from two national, non-profit, peer support based groups: the College Diabetes Network (CDN) and the TuDiabetes Network.

The study aims to 1) develop and pilot and educational video intervention; 2) determine the acceptability and efficiency of various web platforms for engaging college students in completing a survey about their health and alcohol use and to; 3) compare effectiveness of delivery of a brief intervention delivered by a peer versus a provider. The investigators plan to engage 120 college youth with T1D in completing a survey about their health knowledge and alcohol use behaviors.

Baseline survey items will ask participants about knowledge, attitudes, and practices/plans for diabetes self-management and alcohol use in college. In response to survey items, participants will provide information on topics including general and disease-specific health information, as well as attitudes, behavior, beliefs, and knowledge related to alcohol use. Participants will also respond to questions relating to social support, mental health, and perseverance and commitment to long term goals.

Following the baseline survey, participants will be presented with a brief educational video about diabetes self-management and alcohol use risks. Participants will be randomized to receive one of two educational video interventions. One version will be framed and delivered from a peer-based source and the other from a provider, content will otherwise be identical. Participants will receive 2 follow-up surveys; one immediately following viewing the video and the second two weeks later. Both the immediate follow-up and the 2-week follow-up survey will test salience, recall, and effects on health knowledge, beliefs and behavioral intentions.

While the main purpose of the pilot is to ascertain preferences in the absence of preliminary data, our a priori hypothesis is that peer delivery will have greater impact for this population.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be eligible to be included given: self-report of medical diagnosis of Type 1 diabetes, membership in a college diabetes network (CDN) chapter or TuDiabetes (the sampling frame), attendance/matriculation in college, ability to read and understand English (the language of the surveys and the educational vignettes), access to the Internet, ages 17-25 years. Participants must consent to participation in the study and consent to be re-contacted for the two-week follow up assessment, and provide a valid e-mail address for re-contact.

Exclusion Criteria:

* Participants who do not report a diagnosis of T1D, those who are unable to speak/read English at a middle school reading level, use a computer keyboard and/or complete a web-based questionnaire will be excluded. Patients who do not consent to the 2-week follow up or do not provide a valid e-mail address for re-contact will also be excluded.

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 138 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-05-10 (Actual)

PRIMARY OUTCOMES:
Changes in attitudes, beliefs, and intentions about alcohol | Two Weeks
  The primary goal of the proposed project is to determine the effectiveness of diabetes-specific alcohol messaging as delivered by a peer versus a provider, for educating youth in college with Type 1 Diabetes. The ultimate goal is to affect alcohol use behavior, knowledge, attitudes and beliefs and intentions, all of which are proximal to alcohol use behavior. The investigators will assess changes in attitudes, knowledge, beliefs, and intentions about alcohol both immediately following intervention delivery with an immediate follow-up questionnaire, as well with a two-week follow-up questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Elissa R Weitzman, ScD, Principal Investigator — Boston Children's Hospital, Harvard Medical School; Lauren Wisk, PhD, Principal Investigator — Boston Children's Hospital, Harvard Medical School
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wisk LE, Magane KM, Nelson EB, Tsevat RK, Levy S, Weitzman ER. Psychoeducational Messaging to Reduce Alcohol Use for College Students With Type 1 Diabetes: Internet-Delivered Pilot Trial. J Med Internet Res. 2021 Sep 30;23(9):e26418. doi: 10.2196/26418. PMID 34591022
- [Derived] Wisk LE, Nelson EB, Magane KM, Weitzman ER. Clinical Trial Recruitment and Retention of College Students with Type 1 Diabetes via Social Media: An Implementation Case Study. J Diabetes Sci Technol. 2019 May;13(3):445-456. doi: 10.1177/1932296819839503. Epub 2019 Apr 22. PMID 31010315